CLINICAL TRIAL: NCT05330377
Title: Phase Ib Trial of Gilteritinib in Combination With Mitoxantrone, Cladribine, Cytarabine and Filgrastim (GM-CLAG) for Relapsed/Refractory FLT3-mutated Acute Myeloid Leukemia
Brief Title: GM-CLAG in Relapsed/Refractory FLT3-mutated AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Ayman H Qasrawi (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Ayman H Qasrawi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-LEUK-18-PMC
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3; CLAG-M; AML; Relapsed; Refractory; Gilteritinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — gilteritinib; Tablets; Cladribine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Gilteritinib (Dose Level -1: 40 mg/day) (Experimental): Dose escalation for gilteritinib will be conducted according to a BOIN design. Gilteritinib 40 mg/day will be given orally starting day 6 until day 19. CLAG-M chemotherapy will be administered at a fixed dose and schedule as following:
  * Cladribine (CL) 5 mg/m2 I.V. over 2 hours once per day on days 1 to 5, given first.
  * Cytarabine (A) 2,000 mg/m2 I.V. over 4 hours once per day on days 1 to 5, given second, 2 hours after cladribine.
  * Filgrastim (GCSF) 300 mcg S.C. once per day on days 0 to 5, started 24 hours prior to chemotherapy. If WBC is > 20 × 109/L on day 0, the filgrastim dose on day 0 will be omitted.
  * Mitoxantrone (M) 10 mg/m2 I.V. once per day on days 1 to 3
  Interventions: Drug: Gilteritinib 40 MG Oral Tablet; Drug: Cladribine; Drug: Cytarabine; Drug: Filgrastim; Drug: Mitoxantrone
- Gilteritinib (Dose Level 1: 80 mg/day) (Experimental): Dose escalation for gilteritinib will be conducted according to a BOIN design. Gilteritinib 80 mg/day will be given orally starting day 6 until day 19. CLAG-M chemotherapy will be administered at a fixed dose and schedule as following:
  * Cladribine (CL) 5 mg/m2 I.V. over 2 hours once per day on days 1 to 5, given first.
  * Cytarabine (A) 2,000 mg/m2 I.V. over 4 hours once per day on days 1 to 5, given second, 2 hours after cladribine.
  * Filgrastim (GCSF) 300 mcg S.C. once per day on days 0 to 5, started 24 hours prior to chemotherapy. If WBC is > 20 × 109/L on day 0, the filgrastim dose on day 0 will be omitted.
  * Mitoxantrone (M) 10 mg/m2 I.V. once per day on days 1 to 3
  Interventions: Drug: Gilteritinib 40 MG Oral Tablet; Drug: Cladribine; Drug: Cytarabine; Drug: Filgrastim; Drug: Mitoxantrone
- Gilteritinib (Dose Level 2: 120 mg/day) (Experimental): Dose escalation for gilteritinib will be conducted according to a BOIN design. Gilteritinib 120 mg/day will be given orally starting day 6 until day 19. CLAG-M chemotherapy will be administered at a fixed dose and schedule as following:
  * Cladribine (CL) 5 mg/m2 I.V. over 2 hours once per day on days 1 to 5, given first.
  * Cytarabine (A) 2,000 mg/m2 I.V. over 4 hours once per day on days 1 to 5, given second, 2 hours after cladribine.
  * Filgrastim (GCSF) 300 mcg S.C. once per day on days 0 to 5, started 24 hours prior to chemotherapy. If WBC is > 20 × 109/L on day 0, the filgrastim dose on day 0 will be omitted.
  * Mitoxantrone (M) 10 mg/m2 I.V. once per day on days 1 to 3
  Interventions: Drug: Gilteritinib 40 MG Oral Tablet; Drug: Cladribine; Drug: Cytarabine; Drug: Filgrastim; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Gilteritinib 40 MG Oral Tablet — Gilteritinib is an oral FLT3 inhibitor, and is active against both FLT3-ITD and FLT3-TKD mutations. Gilteritinib will be given orally according to the assigned phase I dose cohort starting day 6 until day 19. Participants will be given the daily dose with water as at the same time each morning. Gilteritinib should be taken at least 2 hours after or 1 hour before consuming food.
  Other Names: Xospata
Drug: Cladribine — Cladribine is given intravenously at a dose of 5 mg/m2 I.V. over 2 hours once per day on days 1 to 5.
  Other Names: Leustatin
Drug: Cytarabine — Cytarabine is given intravenously at a dose of 2,000 mg/m2 I.V. over 4 hours once per day on days 1 to 5, given second, 2 hours after cladribine.
  Other Names: cytosine arabinoside (Ara-C)
Drug: Filgrastim — Filgrastim (GCSF) or biosimilar, will be given at a dose of 300 mcg S.C. once per day on days 0 to 5, started 24 hours prior to chemotherapy. If WBC is > 20 × 109/L on day 0, the filgrastim dose on day 0 will be omitted.
  Other Names: GCSF; Filgrastim sndz
Drug: Mitoxantrone — Mitoxantrone is given intravenously at a dose of 10 mg/m2 I.V. over 2 hours once per day on days 1 to 3.
  Other Names: Novantrone

SUMMARY:
The purpose of this study is to evaluate the dose-limiting toxicities (DLT) and define the maximum tolerated dose (MTD) and the recommended phase II study dose of gilteritinib when combined with mitoxantrone, cladribine, cytarabine and filgrastim (GM-CLAG) in participants with FLT3- mutated relapsed or refractory (R/R) acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The treatment of FLT3- mutated relapsed or refractory (R/R) is challenging. Gilteritinib, as a single agent, is the first FLT3 inhibitor to be FDA approved in the R/R setting. This phase I clinical trial will evaluate DLT/MTD and the recommended phase II study dose of gilteritinib when combined with mitoxantrone, cladribine, cytarabine and filgrastim (CLAG-M) in patients with FLT3- mutated R/R AML. This study will also evaluate the pharmacodynamics and pharmacokinetics of gilteritinib when combined with CLAG-M at specific time points. Although this combination has not been established to have superior clinical benefit in comparison to single-agent gilteritinib, the objective of this trial is to provide a possible therapeutic benefit in addition to safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed, morphologically documented AML in first or subsequent relapse or primary induction failure. The diagnosis should be documented within 28 days prior to enrollment.

   1. Relapsed AML is defined as the reappearance of leukemic blasts in the bone marrow, peripheral blood, or any extramedullary site after the attainment of a CR/CRi, detected by morphology, flow cytometry, or immunohistochemistry.
   2. Primary induction failure is defined as failure to achieve a CR or CRi after two courses of induction chemotherapy given per physician's choice or institution's guidelines.
   3. Patients with previous allogeneic hematopoietic stem cell transplantation are allowed to participate, as are prior autologous HCT.
2. Evidence of FLT3-ITD or FLT3-TKD mutations as detected by polymerase chain reaction and/or next-generation sequencing by peripheral blood and/or bone marrow samples obtained at the time of relapse. FLT3 positivity should be documented before enrollment.
3. Allowable prior therapies include: First-line AML therapy including cytarabine, anthracyclines, gemtuzumab ozogamicin, prior hypoemethylating agents with or without venetoclax and/or FLT3 inhibitors.
4. Prior clinical trial participation is allowed with a washout period of experimental drug of at least 4 weeks.
5. Prior treatment with the FLT3 inhibitor gilteritinib is allowed (must be 12 months or greater from time of eligibility screening).
6. Age ≥18 years.
7. ECOG performance status of 0 or 1; Karnofsky 70% or higher (APPENDIX A).
8. Probability of treatment-related mortality (TRM) <13.1% as calculated by performance status, age, platelet count, albumin, secondary vs primary AML, WBC count, creatinine, and percentage of peripheral blood blasts.50

   a. This score corresponds to corresponding to a ≤13.1% probability of 4-week mortality. Although this score was validated for newly diagnosed AML, it was previously used in the relapsed/refractory setting.30,51,52 (see APPENDIX B). An online calculator is available at: https://cstaging.fhcrc-research.org/TRM/).
9. Adequate organ function as defined below:

   1. Creatinine clearance (CrCl) >60 mL/min as measured by Cockcroft-Gault formula (APPENDIX C).
   2. Ejection fraction (EF) ≥ 50% as documented by an echocardiogram or multiple gated cardiac blood pool imaging (MUGA) if the echocardiogram's result is judged to be unreliable by the performing cardiologist.
   3. Total bilirubin ≤ 1.5 × the ULN, unless due to Gilbert's, hemolysis or leukemic infiltration, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, unless caused by leukemic infiltration.
10. Female participants must be either:

    a. Of non-child bearing potential i. postmenopausal status prior to eligibility screening (defined as at least 12 consecutive months of amenorrhea), or ii. undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

    b. Of childbearing potential. These women must agree to all of the following: i. Negative serum/urine pregnancy test at eligibility screening. ii. Abstain from pregnancy during the study and for 6 months after the final study drug administration.

    iii. If heterosexually active, agree to consistently use highly effective contraception per locally accepted standards in addition to a barrier method starting at eligibility screening and throughout the study period and for 6 months after the final study drug administration.
11. Female participants must agree not to breastfeed or donate ova throughout the study drug treatment period and for 6 months after the final study drug administration.
12. Male patients should agree to:

    1. Avoid impregnating a female partner, during the study and for 180 days after the final study drug administration.
    2. Avoid donating sperm during the study and for 180 days after the final study drug administration.
    3. Consistently use highly effective contraception in addition to a barrier method (even if surgically sterilized) along with their partners who are women of childbearing potential, throughout the study drug treatment period and for 6 months after the final study drug administration.
13. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. History of prior treatment with gilteritinib within the last 12 months.
2. Purine analogue (cladribine and fludarabine) treatment as part of their last line of therapy.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gilteritinib or other agents used in this study (CLAG-M).
4. Diagnosis of acute promyelocytic leukemia, BCR/ABL1-positive AML or chronic myelogenous leukemia in blast crisis.
5. Inability to swallow oral medications or gastrointestinal disease limiting absorption of oral agents.
6. Patients with a history of allo-SCT should not have active or acute chronic GVHD requiring systemic immunosuppression; topical GVHD treatment is allowed.
7. Participant has an uncontrolled infection. If a bacterial or viral infection is present, the participant must be receiving definitive therapy and has no signs of progressing infection for 72 hours prior to registration. If a fungal infection is present, the participant must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to registration.

   1. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection.
   2. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
8. Active hepatitis B virus (HBV) infection as evidenced by positive hepatitis B surface antigen and/or Nucleic Acid Amplification Testing (NAAT). Patients with prior history of cleared HBV infection (negative hepatitis B surface antigen, positive hepatitis B surface antibody, and positive hepatitis B core IgG antibody) could be allowed to participate after consultation with a hepatologist, in which case Hep B viral load will be monitored by qPCR per institutional guidelines. In this case, concomitant suppressive antiviral therapy against HBV might be warranted.
9. Uncontrolled HIV infection. Patients who have controlled infection on antiretroviral therapy are allowed, defined as HIV RNA below level of detection for the institution's standard assay.
10. History of heart failure, myocarditis, or cardiomyopathy which requires heart failure directed therapy.
11. Participant has long QT Syndrome at screening.
12. Participant has a Fridericia-corrected QT interval (QTcF) > 450 msec (average of triplicate determinations). Prolonged QTc interval associated with bundle branch block or pacemaking is permitted with written approval of the Principal Investigator (PI).
13. Untreated CNS leukemia. Evaluation of cerebrospinal fluid (CSF) or brain MRI during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening. Patients who previously had CNS leukemia that resolved with therapy should undergo CSF sampling +/- brain MRI within 2 weeks prior to enrollment to exclude CNS relapse.
14. History of auto-immune conditions requiring active immunosuppressive therapy.
15. Patients with uncontrolled intercurrent illness including, but not limited to, symptomatic decompensated congestive heart failure; unstable angina pectoris; cardiac arrhythmia or any acute pulmonary condition requiring need for supplemental oxygen.
16. Participant is receiving concomitant drugs that are strong inducers of CYP3A except for drugs considered essential for the care of the patient.
17. Any medical condition which, in the investigator's opinion, could compromise the patient's safety.
18. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
19. Pregnant or lactating women.
20. Participants who are receiving any other investigational treatment agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) of gilteritinib when combined with mitoxantrone, cladribine, cytarabine and filgrastim (GM-CLAG) | 42 days
  DLT is defined as:
  * Any treatment-related death
  * Grade 4 neutropenia or thrombocytopenia lasting > 42 days from start of cycle in the absence of active AML
    * Any Grade 4 or greater ANC lasting past cycle day 42
    * Any Grade 4 or greater platelets lasting past cycle day 42
  * Grade ≥ 4 organ toxicity (i.e., adverse reactions involving neurologic, pulmonary, cardiac, gastrointestinal, genitourinary, renal, hepatic, or cutaneous systems.)
  * Confirmed Hy's law cases
Maximally Tolerated Dose (MTD) of gilteritinib when combined with mitoxantrone, cladribine, cytarabine and filgrastim (GM-CLAG) | 42 days
  The MTD will be defined as the highest dose of Gilteritinib estimated to have less than 20% hematologic or non-hematologic DLT rates. Enrollment of next patient will be allowed only after prior cohort has completed Cycle 1 and recovered or failure of response has been documented by Day 42.

SECONDARY OUTCOMES:
Complete remission (CR) rate after completing induction chemotherapy with the GM-CLAG combination. | 42 days
  All the following criteria should be met:
  1. bone marrow blasts <5%
  2. absence of circulating blasts and blasts with Auer roda
  3. absence of extramedullary disease
  4. ANC ≥ 1.0 × 109 /L (1000/µL)
  5. platelet count ≥ 100 × 109 /L (100,000/µL).
Complete remission with incomplete hematologic recovery (CRi) after completing induction chemotherapy with the GM-CLAG combination. | 42 days
  All CR criteria should be met except for residual neutropenia ANC ≤ 1.0 × 109 /L (1000/µL) or thrombocytopenia ≤ 100 × 109 /L (100,000 /µL).
Complete remission with partial hematologic recovery (CRh) after completing induction chemotherapy with the GM-CLAG combination. | 42 days
  All CR criteria should be met except for residual neutropenia and thrombocytopenia with at least partial recovery as evidenced by: ANC ≥ 0.5 × 109 /L (500/µL) and platelet count ≥ 50 × 109 /L (100,000/µL).
Composite complete remission (CRc) after completing induction chemotherapy with the GM-CLAG combination. | 42 days
  This is a composite rate of subjects who achieve a CR and those who achieve CRi.
Minimal residual disease status (MRD) after completing induction chemotherapy with the GM-CLAG combination. | Two Induction Cycles (each up to 42 days)
  All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; MRD status will be determined by FLT3 polymerase chain reaction (PCR) testing of bone marrow aspirates obtained at the end of each cycle of induction.
Best response to Induction Therapy | Two Induction Cycles (each up to 42 days)
  Best response is defined as the best measured response (CR, CRp, CRi, or PR) post-treatment.
  Two best responses, up to the time of 2 cycles of treatment period will be defined.
Percentage of patients proceeding to transplantation | Up to 2 years
  To evaluate percentage of patients proceeding to transplantation at anytime during study period
Overall survival (OS) | Up to 2 years
  Defined for all patients of the trial; measured from the date of registration to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Leukemia-free survival (LFS) | Up to 2 years
  Defined only for patients achieving CR, or CRi; measured from the date of achievement of a remission until the date of relapse or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Qasrawi, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No